CLINICAL TRIAL: NCT05130047
Title: A Randomized, Double-Blind, Placebo Controlled Trial of Aldafermin (NGM282) for Treatment of Chronic Diarrhea Due to Bile Acid Malabsorption (BAM)
Brief Title: Aldafermin (NGM282) for Chronic Diarrhea Due to Bile Acid Malabsorption (BAM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Camilleri, MD (Other)
Collaborators: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Michael Camilleri, MD, Professor of Medicine, Pharmacology and Physiology, Atherton and Winifred W. Bean Professor, College of Medicine, Consultant, Division of Gastroenterology and Hepatology., Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-009348
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Chronic Diarrhea; Irritable Bowel Syndrome With Diarrhea; Bile Acid Malabsorption; Bile Acid Diarrhea; Bile Acid Malabsorption Syndrome Type II; Functional Diarrhea
MeSH Terms: interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: 30 participants with diarrhea and laboratory confirmed BAM will be randomized 1:1 to either aldafermin (NGM282), 1 mg, or placebo given daily by subcutaneous injection. Participants and investigators are blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aldafermin (NGM282) (Experimental): Aldafermin (NGM282) is an investigational medication. It is an engineered analog of FGF-19 which reduces synthesis of bile acids and diarrhea caused by elevated bile acids. Participants receive aldafermin (NGM282) 1 mg given by subcutaneous injection once daily for 28 days.
  Interventions: Drug: Aldafermin
- Placebo (Placebo Comparator): A placebo looks exactly like the study drug but contains no active ingredients. It is used to learn if the effects seen are truly from the study drug. Participants receive placebo solution matching aldafermin (NGM282) given by subcutaneous injection once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aldafermin — 1 mg solution
  Other Names: NGM282
  Arms: Aldafermin (NGM282)
Drug: Placebo — Aldafermin placebo solution
  Arms: Placebo

SUMMARY:
This single-center, randomized, double-blind, placebo-controlled study is designed to compare effects of aldafermin, (NGM282), 1 mg, and placebo given daily by subcutaneous injection on bowel functions and hepatic synthesis and fecal excretion of bile acids in patients with diarrhea associated with bile acid malabsorption (BAM).

DETAILED DESCRIPTION:
This single-center, randomized, double-blind, placebo-controlled study is designed to compare effects of aldafermin, NGM282, 1 mg, and placebo given daily by subcutaneous injection on bowel functions and hepatic synthesis and fecal excretion of bile acids in patients with diarrhea associated with bile acid malabsorption (BAM). Thirty patients will receive either aldafermin (NGM282) or placebo, not both. The study includes a 7 to 28-day long prescreen period and a 28-day long treatment period for a maximum study duration of 56 days. Bowel pattern will be assessed by patient-recorded daily bowel pattern diaries. Serum 7-alpha C4 (C4) and fibroblast growth factor 19 (FGF-19) and fecal bile acids will be measured at baseline and Day 14 and Day 28 of treatment. Safety will be assessed through regular monitoring of adverse events, clinical laboratory results, 12-lead ECGs, physical examinations, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, inclusive at Visit 1 Screen.
2. Clinical diagnosis of functional diarrhea or IBS with diarrhea according to Rome III or IV criteria at Visit 1 Screen.
3. Clinical laboratory evidence of BAM (20-22), with at least one of the following results recorded in their past medical history:

   * Serum C4 ≥ 52 ng/mL
   * Fecal BA > 2337 µmoles / 48 hours
   * Total fecal BA > 1000 µmoles / 48 hours + 4 % primary BA
   * Fecal primary BA > 10% / 48 hours
4. Body mass index (BMI) 18.0 to 45.0 kg/m2, inclusive at Visit 1 Screen
5. Understands the study procedures, is willing and able to comply with the study procedures, and is able to give informed consent
6. If treated with any of the following medications, dosing must be stable for 30 days prior to Visit 1 Screen. Patient must agree to maintain the same dose of medication throughout the study:

   * Tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs).
   * Bile acid sequestrants such as colestipol, cholestyramine and colesevelam.
7. Participants must use one highly effective method of contraception for 30 days before the study through 90 days after study completion for males and through 30 days after study completion for females. Highly effective methods of contraception include: Oral, implantable, transdermal or injectable hormonal contraceptives; standard intrauterine device or vaginal ring; Male or female condoms and diaphragms used with spermicide; abstinence from heterosexual intercourse; female partners exclusively sexually active with a surgically sterilized male partner. Females who are surgically sterile having experienced a prior hysterectomy, bilateral salpingectomy, or bilateral oophorectomy or postmenopausal (defined as12 consecutive months with no menses) are not considered to be of childbearing potential.

Exclusion Criteria:

1. Pregnant or lactating
2. Structural or metabolic diseases/conditions that affect the gastrointestinal system
3. Use of the following medications at least 14 days prior to Visit 1 throughout the duration of the treatment period

   * Patients may elect to withdraw from bile acid sequestrants such as colestipol, cholestyramine and colesevelam or they may continue but they must continue at the same dose throughout the study.
   * GI medications including:
   * Anti-nausea agents including trimethobenzamide, promethazine, prochlorperazine, dimenhydrinate, hydroxyzine
   * Osmotic laxative agents including lactulose, sorbitol or PEG solutions as Miralax and Glycolax
   * Prokinetic agents including tegaserod, metoclopramide, prucalopride, domperidone, erythromycin, clarithromycin and azithromycin.
   * 5-HT3 antagonists including alosetron, ondansetron, tropisetron
   * Drugs with a known pharmacological activity at 5-HT4, 5-HT2b or 5-HT3 receptors including tegaserod, ondansetron, granisetron and tropisetron
   * All narcotics including codeine, morphine, and propoxyphene, either alone or in combination
   * Anti-cholinergics including dicyclomine, hyoscyamine, propantheline.
   * Antimuscarinics
   * Tramadol
   * Peppermint oil
   * Systemic antibiotics and antibiotics directed at colonic flora including rifaximin and metronidazole
4. Use of CNS stimulant medications, including methylphenidate, atomoxetine, modafinil, amphetamines or phentermine.
5. Clinically relevant changes in dietary, lifestyle, or exercise regimen within 30 days prior to Visit 1 Screen and throughout the duration of the study
6. Any colonic or major abdominal surgery including bariatric surgery, gastric banding, stomach surgery and intestinal or colonic surgery. Procedures such as appendectomy, cholecystectomy, hysterectomy, caesarean section, or polypectomy are allowed as long as they have occurred at least 3 months prior to Visit 1 Screen.
7. .History of colorectal cancer, inflammatory bowel disease, diverticulitis, ischemic colitis, microscopic colitis or celiac disease
8. History of organic abnormalities of the GI tract, intestinal obstruction, stricture, toxic megacolon, GI perforation, or impaired intestinal circulation.
9. Other GI diseases such as GI bleeding or ulcerations
10. History of cerebrovascular disease including stroke, TIA, acute coronary syndrome, myocardial infarction or unstable angina
11. Clinically significant cardiac history or presence of electrocardiogram (ECG) findings at Visit 1 Screen:

    * Abnormal heart rate < 40 or > 100 beats per minute
    * QTc interval > 470 milliseconds (ms)
    * QRS interval ≥ 110 ms
    * PR interval ≥ 220 ms
12. Hepatic dysfunction including abnormal serum alanine aminotransferase [ALT] or aspartate transaminase [AST] > 3 × upper limit of normal [ULN]); total direct bilirubin > 2 × ULN, or alkaline phosphatase > 2 × ULN at Visit 1 Screen
13. Clinically significant renal insufficiency including serum creatinine > 2.5 mg/dL at Visit 1 Screen
14. History of severe head injury or history of seizures
15. History of suicide attempt or a hospitalization for a major psychiatric condition within 1 year prior to Visit 1 Screen. At Visit 1 Screen or during the optional remote consent and eligibility review, participants will complete the Hospital Anxiety and Depression questionnaire. If either score for anxiety or depression individually exceeds 8, the score will be discussed. The patient will be and advised whether to participate or whether to see their primary care physician.
16. History of alcohol use disorder or substance use disorder within 2 years of Visit 1 Screen.
17. Significant history or clinical manifestation of any endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, GI, neurological or psychiatric disorder, malignancy (with the exception of treated basal cell carcinomas), or any other condition that would prevent the individual from participating in the study due to risk to the scientific validity of study assessments or to personal well-being of the patient.
18. Participated in another clinical study that includes an investigational drug or a biologic therapy within 30 days or 5 half-lives, whichever time period is longer, prior to Visit 1 Screen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Aldafermin (NGM282): Aldafermin (NGM282) is an investigational medication. It is an engineered analog of FGF-19 which reduces synthesis of bile acids and diarrhea caused by elevated bile acids. Participants received aldafermin (NGM282) 1 mg given by subcutaneous injection once daily for 28 days.
  Aldafermin: 1 mg solution
- Placebo: A placebo looks exactly like the study drug but contains no active ingredients. It is used to learn if the effects seen are truly from the study drug. Participants received placebo solution matching aldafermin (NGM282) given by subcutaneous injection once daily for 28 days.
  Placebo: Aldafermin placebo solution
Period: Overall Study
Arm/Group | Aldafermin (NGM282) | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aldafermin (NGM282) | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.0 [40.0 to 53.0] | 43.0 [39.0 to 58.0] | 43.0 [40.0 to 53.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Fasting Serum C4 Levels
Description: Fasting serum C4 is measured by liquid chromatography-mass spectrometry.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: ng/ML
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
ng/ML | 2.2 [1.6 to 3.3] | 50.4 [25.8 to 106.0]

2. Primary Outcome: Change in Stool Consistency From Baseline to Day 28
Description: Stool consistency as reported by the patient in daily bowel pattern diaries. Stool consistency is based on Bristol Stool Form Scale (BSFS) 1: Hard lumps; 2:Lumpy sausage; 3: Cracked sausage; 4: Smooth sausage; 5: Soft lumps; 6: Mushy; 7: Watery. spectrometry.
Time Frame: Baseline, 28 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | -0.4 [-1.2 to 0.1] | -0.02 [-0.4 to 0.3]

3. Secondary Outcome: Stool Consistency
Description: Stool consistency as reported by the patient in daily bowel pattern diaries. Stool consistency is based on Bristol Stool Form Scale (BSFS) 1: Hard lumps; 2:Lumpy sausage; 3: Cracked sausage; 4: Smooth sausage; 5: Soft lumps; 6: Mushy; 7: Watery.
Time Frame: 14 days, 28 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale
  Day 14 | 4.6 [4.3 to 5.0] | 4.8 [4.0 to 5.3]
  Day 28 | 4.4 [4.2 to 5.0] | 5.1 [4.4 to 5.5]

4. Secondary Outcome: Abdominal Pain Score
Description: Abdominal pain rated by patient using an 11-point scale, 0 to 10 inclusive with 0 as none and 10 as worst imaginable abdominal pain.
Time Frame: baseline, 28 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 0.9 [0.0 to 3.6] | 0.4 [0 to 1.0]
  Day 28 | 0.6 [0.0 to 1.3] | 0.5 [0.1 to 1.1]

5. Secondary Outcome: Bowel Movements
Description: The total number of bowel movements per day reported by the participant in the daily bowel pattern diary.
Time Frame: baseline, 28 days
Measure: Median (Inter-Quartile Range); unit: bowel movements per day
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
bowel movements per day
  Baseline | 2.3 [1.9 to 3.2] | 2.3 [1.8 to 3.0]
  Day 28 | 2.3 [2.1 to 3.6] | 2.1 [1.7 to 2.7]

6. Secondary Outcome: Proportion of Fecal Secretory (CDCA + DCA) Bile Acid as Measured in a Random Stool Sample by a Validated Laboratory Assay.
Description: Fecal secretory bile acids are expressed as a percentage of the total bile acids as measured by high performance liquid chromatography-mass spectrometry.
Time Frame: Baseline, 14 days, 28 days
Measure: Median (Inter-Quartile Range); unit: percentage of the total bile acids
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
percentage of the total bile acids
  Baseline | 63.8 [58.3 to 66.7] | 63.2 [57.4 to 66.6]
  Day 14 | 43.2 [32.5 to 53.5] | 59.2 [53.1 to 63.9]
  Day 28 | 45.5 [39.8 to 55.6] | 60.0 [46.3 to 65.1]

7. Secondary Outcome: Proportion of Fecal Primary (CDCA + CA) Bile Acid as Measured in a Random Stool Sample by a Validated Laboratory Assay.
Description: Fecal primary bile acids are expressed as a percentage of the total bile acids as measured by high performance liquid chromatography-mass spectrometry.
Time Frame: Baseline,14 days, 28 days
Measure: Median (Inter-Quartile Range); unit: percentage of the total bile acids
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
percentage of the total bile acids
  Baseline | 5.4 [1.9 to 14.6] | 5.2 [2.0 to 12.9]
  Day 14 | 10.3 [3.3 to 15.4] | 2.8 [0.7 to 9.8]
  Day 28 | 9.9 [3.0 to 20.0] | 14.3 [7.4 to 27.4]

8. Secondary Outcome: Total Fecal Bile Acid Concentration in a Random Stool Sample as Measured by a Validated Laboratory Assay.
Description: Total fecal bile acids concentration in micromoles of bile acid per gram stool as measured by high performance liquid chromatography-mass spectrometry.
Time Frame: baseline,14 days, 28 days
Measure: Median (Inter-Quartile Range); unit: mmol/g
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 15 | 15
mmol/g
  Baseline | 3.1 [1.9 to 4.0] | 3.5 [1.9 to 4.3]
  Day 14 | 0.5 [0.3 to 0.7] | 2.7 [1.2 to 5.1]
  Day 28 | 0.5 [0.3 to 0.8] | 3.6 [1.0 to 7.3]

9. Secondary Outcome: Total Aldafermin Concentration in Serum as Measured by a Validated Laboratory Assay
Description: Validated aldafermin concentration (PK) laboratory assay
Time Frame: baseline, 14 days, 28 days
Population: Data was not collected nor analyzed
Arm/Group | Aldafermin (NGM282) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study for each participant, approximately 28 days
Arm/Group | Aldafermin (NGM282) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 14/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldafermin (NGM282) (N=15) | Placebo (N=15)
Myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aldafermin (NGM282) (N=15) | Placebo (N=15)
Increased diarrhea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Other gastrointestinal symptoms (Gastrointestinal disorders) | 3 | 3
Increased LDL Cholesterol (Investigations) | 4 | 0
Irritation at injection site (Skin and subcutaneous tissue disorders) | 3 | 1
Infections (Infections and infestations) | 5 | 2
Headache (Nervous system disorders) | 2 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 | 2
Metabolism and Nutrition (Metabolism and nutrition disorders) | 2 | 0
Reanl and urinary (Renal and urinary disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT05130047/Prot_SAP_000.pdf